CLINICAL TRIAL: NCT02995642
Title: Targeted PET/CT and PET/MRI Imaging of Vascular Inflammation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Resources not secured
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Andrei Iagaru, Associate Professor of Radiology (Nuclear Medicine) at the Stanford University Medical Center, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 26885
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Aortic Aneurysm, Abdominal; Carotid Atherosclerosis
Keywords: Aortic Aneurysm, Abdominal; Carotid Stenosis; Atherosclerosis; Angiogenesis; Inflammation; Macrophages; Positron-Emission Tomography; Computerized tomography; Magnetic Resonance Imaging; (18F)FPP(RGD)2
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Carotid Artery Diseases; Carotid Stenosis; Atherosclerosis; Inflammation | interventions — FPP(RGD)2; Positron-Emission Tomography; Tomography, Emission-Computed; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-FPPRGD2 (Experimental): Subjects (with either carotid atherosclerosis stenosis or AAA) will receive a single intravenous injection of 10mCi of 18F-FPPRGD2 and will undergo positron emission tomography/computed tomography (PET/CT) or PET/MRI (PET/magnetic resonance imaging) imaging 45-60 minutes after injection.
  Interventions: Drug: 18F-FPPRGD2; Device: Positron emission tomography; Procedure: Computed tomography; Device: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: 18F-FPPRGD2 — One single intravenous injection.
  Other Names: Fluorine-18-labeled RGD peptide [18F] FPA-PEG3-E[c(RGDyK)]2
Device: Positron emission tomography — Undergo 18F-FPPRGD2 PET/CT or PET/MRI
  Other Names: PET; PET scan; tomography, emission computed
Procedure: Computed tomography — Undergo 18F-FPPRGD2 PET/CT or PET/MRI
  Other Names: tomography, computed
Device: Magnetic Resonance Imaging — Undergo 18F-FPPRGD2 PET/CT or PET/MRI
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging

SUMMARY:
Stroke and abdominal aortic aneurysms (AAAs) are common and highly lethal vascular diseases. Angiogenesis and infiltration of inflammatory cells such as macrophages may cause stroke and AAAs.

The purpose of this study is to test PET/CT and PET/MRI imaging to specifically detect those diseases using a new developed agent (18F-FPPRGD2) that can target angiogenesis and macrophages.

DETAILED DESCRIPTION:
20 subjects with either carotid bifurcation stenosis of >50% by ultrasound on at least one side (10 patients) or advanced AAAs (10 patients) and surgical intervention planned will be identified from physicians from the Division of Vascular Surgery at Stanford.

Either a PET/CT or a PET/MRI will be performed for each subject:

* PET/CT scans will be performed in 3D mode using GE Discovery 600 or GE Discovery 690 scanners (GE Healthcare).
* PET/MRI scans will be performed using the novel PET/MRI system at Stanford, including a sensitive PET time-of-flight (TOF) scanner with an advanced 3T MRI scanner.

The study patients will receive an intravenous administration of 10mCi of the prescribed radiotracer (18F-FPPRGD2). PET/CT or PET/MRI images will be obtained starting 45-60 minutes after radiotracer administration. For PET/CT, each image acquisition will begin with a non-contrast CT scan obtained from the vertex through the mid-thighs of the subjects. For PET/MRI, non-contrast images of the carotid or aorta will be performed. PET imaging will follow. Patient's vital signs will be monitored during the procedure and a physician will be available if there is need for immediate medical attention. The PET images will be reconstructed with a standard iterative algorithm using GE software release 5.0.

After the planned surgery, we will also assess the histopathological correlation between the disease lesions and PET/CT or PET/MRI imaging characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 year-old at the time of radiotracer administration
* Provides written informed consent
* Patients diagnosed with either carotid artery stenosis or abdominal aortic aneurysms (AAAs) as identified in Vascular Surgery, in whom a surgical procedure is scheduled
* Able to remain still for duration of an imaging procedure (about one hour).

Exclusion Criteria:

* Less than 18 year-old at the time of radiotracer administration
* Unable to provide written informed consent
* Pregnant women
* Prior carotid or abdominal surgery
* History of radiation therapy to the neck and abdomen
* MRI contraindications (including ferromagnetic objects or devices).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
SUVmax of 18F-FPPRGD2 uptake by lesions (carotid atherosclerotic plaque or AAA). | Up to 60 minutes post-injection (at time of scan)
  The arterial standardized uptake value (SUV) for carotid plaque or AAA will be calculated as the mean pixel activity within the region of interest (ROI).
  By averaging the SUV values for each artery slice, we will derived a mean SUV value for the entire artery (arterial SUV). This will be corrected for blood activity by division by the average blood SUV estimated from either the inferior vena cava or jugular vein to produce a blood-corrected artery SUV, known as the arterial tissue-to-background ratio (TBR).
Percent agreement of 18F-FPPRGD2 PET with pathology | Up to 60 minutes post-injection (at time of scan)
  After the planned surgical procedure, the accuracy of 18F-FPPRGD2 PET as percent agreement with pathology (including angiogenesis and inflammation assessment) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Michael V. McConnell, MD, MSEE, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mittra ES, Goris ML, Iagaru AH, Kardan A, Burton L, Berganos R, Chang E, Liu S, Shen B, Chin FT, Chen X, Gambhir SS. Pilot pharmacokinetic and dosimetric studies of (18)F-FPPRGD2: a PET radiopharmaceutical agent for imaging alpha(v)beta(3) integrin levels. Radiology. 2011 Jul;260(1):182-91. doi: 10.1148/radiol.11101139. Epub 2011 Apr 18. PMID 21502381
- [Background] Kitagawa T, Kosuge H, Chang E, James ML, Yamamoto T, Shen B, Chin FT, Gambhir SS, Dalman RL, McConnell MV. Integrin-targeted molecular imaging of experimental abdominal aortic aneurysms by (18)F-labeled Arg-Gly-Asp positron-emission tomography. Circ Cardiovasc Imaging. 2013 Nov;6(6):950-6. doi: 10.1161/CIRCIMAGING.113.000234. Epub 2013 Aug 30. PMID 23995363